CLINICAL TRIAL: NCT05069558
Title: Prospective Randomized Multi-center Controlled Clinical Investigation Comparing Patent Foramen Ovale (PFO) Outcomes of the Occlutech Flex II PFO Occluder to Standard of Care PFO Occlusion
Brief Title: Comparing PFO Outcomes of the Occlutech Flex II PFO Occluder to Standard of Care PFO Occlusion
Acronym: OCCLUFLEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCC2021_02
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Patent Foramen Ovale; PFO
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational PFO Closure Device (Experimental): PFO closure with the study Occlutech Flex II PFO device.
  Interventions: Device: Investigational PFO Closure Device
- Standard of Care PFO Closure Device (Active Comparator): PFO closure with either of the standard of care PFO occlusion devices; Amplatzer PFO Occluder or the Gore Cardioform PFO Occluder.
  Interventions: Device: Standard of Care PFO Closure Device

INTERVENTIONS:
Device: Investigational PFO Closure Device — Occlutech Flex II PFO Closure Device
  Arms: Investigational PFO Closure Device
Device: Standard of Care PFO Closure Device — Amplatzer PFO Occluder and Gore Cardioform PFO Occluder
  Arms: Standard of Care PFO Closure Device

SUMMARY:
The objective of this study is to investigate whether percutaneous PFO closure with the Occlutech Flex II PFO Occluder is non-inferior to the AMPLATZER™ PFO Occluder and Gore® Cardioform Septal Occluder in closure of the PFO, prevention of recurrent embolic stroke, and device/procedure related Serious Adverse Events (SAE).

ELIGIBILITY:
Inclusion Criteria: Subjects with a PFO and cryptogenic stroke:

* PFO defined as visualization of microbubbles (during Trans Esophageal Echo (TEE)) in the left atrium within three cardiac cycles of right atrial opacification at rest and/or with Valsalva.
* Cryptogenic stroke defined as a stroke of unknown cause.
* Stroke defined as an acute focal neurological deficit, presumed to be due to focal ischemia, and either:
* Symptoms persisting ≥24 hours OR
* Symptoms persisting <24 hours with Magnetic Resonance Imaging (MRI) or Computer Tomography (CT) findings of a new, neuroanatomically relevant, cerebral infarct.

Exclusion Criteria:

* Age < 18 years
* Myocardial Infarction (MI) or unstable angina within 6 months.
* Severe mitral valve stenosis, severe aortic valve stenosis, or severe regurgitation.
* Left Ventricle Ejection Fraction (LVEF) <35%.
* Uncontrolled hypertension or diabetes mellitus despite medications.
* Subjects contraindicated for aspirin or clopidogrel.
* Presence of other comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical trial or to comply with follow up requirements, or impact the scientific soundness of the clinical trial results.
* Qualifying stroke with Modified Rankin score >3.
* Anatomy in which the device would interfere with intracardiac or vascular structures.
* Life expectancy < 2 years.
* Participation in another clinical study that can interfere with the results of this study
* Exclusion for patients with known causes of ischemic stroke:
* Atrial fibrillation/atrial flutter (chronic or intermittent).
* Left Ventricle (LV) aneurysm, intracardiac thrombus, or tumor.
* Mitral or aortic valve vegetation or prosthesis.
* Aortic arch plaques protruding >4 mm into the lumen.
* Atherosclerosis or arteriopathy of intra- or extracranial vessels with >50% diameter stenosis in the artery supplying the infarcted territory.
* Another cause of right-to-left shunting (e.g., an Atrial Septal Defect (ASD) or a fenestrated atrial septum).
* Presence of an arterial hypercoagulable state.
* Lacunar infarct probably due to intrinsic small vessel as the qualifying event, defined as an ischemic stroke in the distribution of a single, small deep penetrating vessel in a patient with any of the following:
* A history of hypertension (except in the first week post stroke).
* A history of diabetes mellitus.
* Age ≥50 years.
* MRI or CT with leukoaraiosis greater than symmetric, well-defined periventricular caps, or bands (European Task Force on Age-Related White Matter Changes rating scale score >0).
* Arterial dissection as the qualifying event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Effective Closure Rate of PFO | Twelve Months

SECONDARY OUTCOMES:
Non-Fatal Recurrent Stroke | Enrollment to 12 Months

OTHER OUTCOMES:
Safety: Device and Procedure Related Serious Adverse Events | Enrollment to Twelve Months, Annually thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: David Thaler, MD, PhD, FAHA, Study Chair — Tufts Medical Center and Tufts University School of Medicine; Steven Yakubov, MD, FACC, MSCAI, Study Chair — OhioHealth Heart & Vascular
Locations (48):
- United States (27):
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Stanford University Medical Center, Stanford, California
  - Los Robles Medical Center, Thousand Oaks, California
  - Colorado Heart and Vascular PC / St. Anthony Hospital, Lakewood, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Louisville, Louisville, Kentucky
  - MaineHealth, Portland, Maine
  - Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Essentia Health, Duluth, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Valley Hospital, Paramus, New Jersey
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
- Canada (6):
  - University of Alberta Mazankowski Heart Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montreal (CHUM), Montreal, Quebec
  - Institut de Cardiologie de Montréal, Montreal, Quebec
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Copenhagen, Copenhagen
- Heart and Lung Center, Helsinki University Hospital, Helsinki, Finland
- France (3):
  - CHU Grenoble Alpes, La Tronche
  - Hôpital Privé Jacques Cartier, Massy
  - CHU Toulouse Rangueil, Toulouse
- Germany (5):
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Asklepios Klinik Altona Hamburg, Hamburg, Hamburg
  - CardioVasculäre Centrum Frankfurt, Frankfurt
  - Universitätsklinik Heidelberg, Heidelberg
  - University Heart Center Lübeck, Lübeck
- Netherlands (2):
  - Amsterdam University Medical Center, Amsterdam
  - Erasmus University Medical Centre, Rotterdam
- United Kingdom (2):
  - University Hospitals Sussex, Brighton, East Sussex
  - Royal Victoria Hospital, Belfast

IPD SHARING:
Plan to Share IPD: No